CLINICAL TRIAL: NCT04384900
Title: Accelerated Prone Position Ventilation of Patients With COVID-19
Acronym: PROVENT-COVID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigators
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-20027361
Record Dates: First submitted 2020-05-11; First posted 2020-05-12 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Prone position ventilation; ARDS; intensive care unit; respiratory failure
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated prone position (Experimental): Prone position ventilation initiated as soon as possible following intubation. The patients are maintained in a prone position for 12-16 hrs daily for 5 days, unless one of the following criteria are met: Substantial improvement and/or imminent extubation, Worsening oxygenation with prone position, Serious Adverse Reactions (SARs) occurring during a prone session and leading to its immediate interruption. Following the five day intervention period, prone position ventilation will be continued according to the intervention in the control group
  Interventions: Procedure: Prone position ventilation
- Standard prone position (Active Comparator): Standard of care: Prone position applied according to standard indications (severe ARDS not improving with 12-24 hours of mechanical ventilation with PaO2-to-FiO2 ratio (PAF) < 150 mmHg with FiO2 of ≥0.6, a positive end-expiratory pressure (PEEP) of ≥5 cm of water, and a tidal volume of about 6 ml per kilogram of predicted body weight). Until one of the following are met: Substantial improvement and/or imminent extubation, Worsening oxygenation with prone position, Serious Adverse Reactions (SARs) occurring during a prone session and leading to its immediate interruption.
  Interventions: Procedure: Prone position ventilation

INTERVENTIONS:
Procedure: Prone position ventilation — Patients are placed in a prone position using specialized equipment.

SUMMARY:
Prone position ventilation is frequently used in the ICU to treat severe hypoxemia in patients with COVID-19 associated acute respiratory distress syndrome (ARDS). The aim of the PROVENT-COVID study is to assess whether applying prone position ventilation immediately after intubation reduces the duration of mechanical ventilation compared to prone position ventilation according to standard criteria for prone position.

DETAILED DESCRIPTION:
In patients with COVID-19 the incidence of ARDS is 15% and the all-cause mortality 4%. No treatment has been shown to improve the outcome of these patients.

Mechanical ventilation in the prone position decreases mortality with around 50% when applied to patients with severe respiratory failure. Applying prone position earlier in patients with COVID-19 could have several benefits, but may also carry significant side-effects and an increased workload for the health-care personnel. It is urgently needed to assess whether this potential life-saving intervention is effective.

The aim of the PROVENT-COVID is to determine whether prone position ventilation, initiated immediately after intubation, lead to more days alive without respiratory support compared to prone position initiated according to standard indication in patients with COVID-19 associated respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Admitted to an intensive care unit.
* Indication for intubation and mechanical ventilation
* No suspicion of significant cardiac failure induced pulmonary edema.
* Suspected COVID-19 or positive SARS-Cov-2 PCR or equivalent diagnostic test.
* Inclusion as soon as possible and maximum 12 hours after intubation.

Exclusion Criteria:

* Contraindication for prone position ventilation: Suspected high intracranial pressure, massive hemoptysis requiring an immediate surgical or interventional radiology procedure, tracheal surgery or sternotomy during the previous 15 days, serious facial trauma or facial surgery during the previous 15 days, cardiac pacemaker inserted in the last 2 days, unstable spine, femur, or pelvic fractures, single anterior chest tube with air leaks, body constitution that is incompatible with prone position ventilation (i.e. high BMI)
* Admitted under duress (psychiatry).
* Pregnant or breastfeeding.
* Mechanical ventilation in prone position prior to inclusion in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Days alive without respiratory life support (invasive mechanical ventilation) at day 28. | 28 days after randomization
  Number of days where patients are alive and not receiving mechanical ventilation

SECONDARY OUTCOMES:
Days alive and out of hospital on day 28 after randomisation. | 28 days
  Number of days alive and out of hospital
Days alive at day 28 without life support (vasopressor/inotropic support, invasive mechanical ventilation or renal replacement therapy). | 28 days
  Number of days where patients are alive and not receiving life support
Number of participants with one or more SARs as described in section 6.1 plus incidence of new persistent nerve injury or grade 3 or 4 (full-thickness skin loss or worse) pressure wounds. | 28 days
  Number of patients with severe adverse reaction
28-days all-cause mortality. | 28 days
  Number patients who have died

CONTACTS AND LOCATIONS:
Overall Officials: Morten H Bestle, MD, PhD, Principal Investigator — Nordsjællands Hospital, University of Copenhagen
Locations (1):
- Nordsjællands Hospital, Hillerød, Region Hovedstanden, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available 9 months after the publication of the outcome data according to the recent ICMJE recommendations
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 9 months after publication of primary results